CLINICAL TRIAL: NCT07286630
Title: Prevalence Of Disability And Fear Avoidance Beliefs Among Egyptian Physical Therapists With Chronic Non Specific Low Back Pain
Brief Title: Prevalence Of Disability And Fear Avoidance Beliefs
Status: Enrolling by invitation | Type: Observational
Sponsor: Dina Abdelhady Hammad Attia Ahmed (Other)
Responsible Party: Sponsor-Investigator, Dina Abdelhady Hammad Attia Ahmed, Principal investigator, Cairo University
Organization: Cairo University (Other)
Other Study IDs: PDAF
Record Dates: First submitted 2025-09-22; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Chronic Non-specific Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fear avoidance beliefs questionnaire — * Fear avoidance beliefs will be measured using the FABQ. It contains 16 items, scored from 0-6 (completely agree to completely disagree). It consists of two subscales, the physical activity subscale (FABQ PA), scored out of 24 (scores of ≤15 indicate low and >15 indicate high fear avoidance), and work (FABQ W), scored out of 42 points (scores of ≤34 indicate low and >34 indicate high fear avoidance)
  * Oswestrydisability examines the level of disability in 10 everyday activities of daily living.
  * Pain intensity -Personal care -Lifting
  * Walking -Sitting -Standing
  * Sleeping -Sex (if applicable)
  * Social -Travel (Physiopedia, n.d.).
  * Each component is assigned a value between 0 and 5, with 5 indicating the most disability. The index is calculated by dividing the total score by the range of scores and multiplying the result by 100 to get the index's percentage value .

SUMMARY:
Three hundred eighty -one egyptian physical therapists of both genders with age 25-55 years old in Cairo governorate who have worked for at least two years.The study will be conducted to investigate the prevalence of disability and fear avoidance beliefs among egyptian physical therapists with chronic non-specific low back pain (CNSLBP), and data will be collected through self-administered questionnaires distributed electronically.Participants were recruited from various public and private physical therapy centers and hospitals in Cairo .

DETAILED DESCRIPTION:
1. Sujects:

   Three hundred eighty -one egyptian physical therapists of both genders with age 25-55 years old in Cairo governorate who have worked for at least two years.The study will be conducted to investigate the prevalence of disability and fear avoidance beliefs among egyptian physical therapists with chronic non-specific low back pain (CNSLBP) , and BMI 18:30 kg/m2 and data will be collected through self-administered questionnaires distributed electronically.Participants were recruited from various public and private physical therapy centers and hospitals in Cairo .
2. Instrumentation for assessment:

Patients will be assessed by:

1. Fear-Avoidance Beliefs Questionnaire ( FABQ ) for assessing fear-avoidance beliefs in individuals with low back pain
2. Oswestry Disability Index (ODI) for measurement of disability in patients with low back pain

Assessment procedures:

This study will include 381 subjects both male and female physical therapists who have worked for at least two years. The assessment will be performed one time for each participant by the same physiotherapist. All participants will first be checked to see if they are matching the inclusion and exclusion criteria after that they will inform consent.

A pretested, self-administered, structured questionnaire will be used for data collection. The survey examined demographic data, gender, age, weight, height, smoking habits, drinking habits, marital status, history of LBP in the last year, the duration of the last LBP, pain consultation at a hospital, history of LBP treatment in the last year, current occupation, history of heavy physical labor, duration of driving or riding, history of exercise, duration of sitting, and duration of standing .

1. The Fear avidance beliefs Questionnaire (FABQ): will be sent to physical therapists working in Cairo. Participants will be selected from public and private physical therapy clinics in Cairo. Responses will be collected by an electronic survey tool (i.e.,Google Form) and exported for statistical analysis with SPSS.

   -Fear avoidance beliefs will be measured using the FABQ. It contains 16 items, scored from 0-6 (completely agree to completely disagree). It consists of two subscales, the physical activity subscale (FABQ PA), scored out of 24 (scores of ≤15 indicate low and >15 indicate high fear avoidance), and work (FABQ W), scored out of 42 points (scores of ≤34 indicate low and >34 indicate high fear avoidance) .
2. Oswestry Disability Index (ODI): The ODI will be used to assess the functional disability in NSCLBP.

   * The questionnaire examines the level of disability in 10 everyday activities of daily living.
   * Pain intensity -Personal care -Lifting
   * Walking -Sitting -Standing
   * Sleeping -Sex (if applicable)
   * Social -Travel
   * Each component is assigned a value between 0 and 5, with 5 indicating the most disability. The index is calculated by dividing the total score by the range of scores and multiplying the result by 100 to get the index's percentage value .
   * Scores are calculated as follows: [total score/(5 x number of questions answered)] x 100% (Shirley Ryan AbilityLab, n.d.).
   * Interpretation:
   * Functional disability will be classified into the following five classes:
   * minimal disability (0-20)
   * moderate disability (21-40)
   * severe disability (1-60)
   * crippled (61-80); and
   * being bed-bound (81-100)

ELIGIBILITY:
Inclusion Criteria:

* Male and female Egyptian physical therapists who have worked for at least two years.
* Working age from 25 to 55 years .
* Those experiencing localized pain from the lower margin of the twelfth rib to the lower gluteal folds for more than three months were included in the NS-CLBP .
* Physical therapists who are fluent in English language.
* BMI 18:30 kg/m2 .

Exclusion Criteria:

* Participants with a history of orthopaedic spine disease or surgery were excluded .
* cauda equina lesion, malignancy, infection, history of spinal surgeries, pregnancy, pain related to mensuration, and mental illness.

Ages: 25 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: This study will target the egyptian physical therapists in Cairo governorate who have worked for at least two years. This cross-sectional study included a convenience sample of Egyptian physical therapists diagnosed with chronic non-specific low back pain (CNSLBP). Participants were recruited from various public and private physical therapy centers and hospitals in Cairo .
Sampling Method: Non-Probability Sample
Enrollment: 381 (Estimated)
Dates: Start 2025-09-07 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Disaility Among Egyptian Physical Therapists With Chronic Non Specific Low Back Pain | 1 month
  * Fear avoidance beliefs will be measured using the FABQ. It contains 16 items, scored from 0-6 (completely agree to completely disagree). It consists of two subscales, the physical activity subscale (FABQ PA), scored out of 24 (scores of ≤15 indicate low and >15 indicate high fear avoidance), and work (FABQ W), scored out of 42 points (scores of ≤34 indicate low and >34 indicate high fear avoidance)
  * Oswestrydisability examines the level of disability in 10 everyday activities of daily living. -Pain intensity -Personal care -Lifting -Walking -Sitting -Standing -Sleeping -Sex (if applicable) -Social -Travel (Physiopedia, n.d.). -Each component is assigned a value between 0 and 5, with 5 indicating the most disability. The index is calculated by dividing the total score by the range of scores and multiplying the result by 100 to get the index's percentage value .

CONTACTS AND LOCATIONS:
Overall Officials: Dina Abdelhady Hammad, Bachaleor, Principal Investigator — Cairo University
Locations (1):
- Faculty of physical therapy, Cairo, Egypt